CLINICAL TRIAL: NCT03037073
Title: Impact of Duloxetine on Succinylcholine-induced Postoperative Myalgia During Direct Microlaryngoscopic Surgeries: Randomized Controlled Double-blind Study
Brief Title: Duloxetine for Succinylcholine-induced Postoperative Myalgia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed F. Mostafa, Lecturer of Anesthesia and Intensive Care, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Duloxetine POM
Record Dates: First submitted 2017-01-26; First posted 2017-01-31 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Postoperative Myalgia
Keywords: Duloxetine; Succinylcholine; Postoperative Myalgia; Microlaryngoscopy
MeSH Terms: interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group D (Active Comparator): 35 patients will receive duloxetine (Cymbalta; Eli Lilly & Company, Indiana, USA) 30 mg orally with sips of water, 2 h before induction of anesthesia.
  Interventions: Drug: Duloxetine
- Group C (Active Comparator): 35 patients will receive similar-looking placebo capsules (starch capsules) orally with sips of water, 2 h before induction of anesthesia.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Duloxetine — 35 patients will receive duloxetine (Cymbalta; Eli Lilly & Company, Indiana, USA) 30 mg orally with sips of water, 2 h before induction of anesthesia.
  Arms: Group D
Drug: Placebo oral capsule — 35 patients will receive similar-looking placebo capsules (starch capsules) orally with sips of water, 2 h before induction of anesthesia.
  Arms: Group C

SUMMARY:
For >60 years, succinylcholine is still being administered as a selective relaxant for rapid sequence intubation by anesthesiologists in many countries. It has been shown to possess unique features such as low cost, fast-acting, short half-life, safe metabolites, and causing excellent muscle relaxation for intubation. It has many side effects as well. Postoperative myalgia (POM), with an incidence rate of ~41%-92%, is one of the most common side effects of this drug and can take several days to cause significant discomfort in patients. However, its effect is felt more in the throat, neck, shoulder, and abdominal muscles and is common among patients with outpatient surgery. Due to its unknown real context of pathogenesis and in an effort to reduce the incidence and severity of succinylcholine-induced myalgia, various medications including nondepolarizing muscle relaxants, benzodiazepines, magnesium sulfate, opioids, gabapentin, and nonsteroidal anti-inflammatory drugs have been tested, with varying degrees of success.

Duloxetine is an US Food and Drug Administration-approved analgesic used for various pain syndromes, including diabetic peripheral neuropathy and fibromyalgia. The underlying mechanism for duloxetine against these pain syndromes remains unclear, but it may involve three major central nervous system (CNS) targets: (1) serotonin transporter (Ki, 4.6 nM), (2) norepinephrine transporter (Ki, 16 nM), and (3) dopamine transporter (Ki, 370 nM). In the past, the antidepressant action was often thought to be the primary mechanism for its analgesic efficacy. This theory was addressed later by "Path Analysis," and the result showed that duloxetine affects pain directly rather than indirectly through mood improvement. In addition to these multiple CNS targets, duloxetine, like the antidepressant amitriptyline and the local anesthetic bupivacaine, blocks voltage-gated Na+ channels. Because neuronal Na+ channels are present in both CNS and peripheral nervous systems, such a finding expands the possible analgesic action and locus of duloxetine.

DETAILED DESCRIPTION:
Eligibility and type of the study: This prospective randomized placebo-controlled double-blind study will be conducted after approval from the Institutional Ethics Committee and obtaining written informed consent from patients undergoing elective direct microlaryngoscopic surgeries under general anesthesia.

Sample size: Sample size calculation is based on the pilot study, where the incidence of POM in outpatient cases is found to be more than 70% and intervention that can cause 25% reduction in incidence of POM will be interesting. With a power of 90% and type I error of 5%, 32 patients will be required in each group (α=0.05 and β=90%), but to avoid possible loss of samples (dropouts) during the study, the number of patients in each group will be increased to 35 to be a total of 70 patients.

Patients: Seventy patients will be enrolled in this study. They will be equally divided into two groups. Group D (duloxetine group): 35 patients will receive duloxetine (Cymbalta; Eli Lilly & Company, Indiana, USA) 30 mg orally with sips of water, 2 h before induction of anesthesia. Group C (control group) 35 patients will receive similar-looking placebo capsules (starch capsules) orally with sips of water, 2 h before induction of anesthesia.

Anesthetic Technique and Data Collection: The patients will not be pre-medicated. The study drugs will be given to patients by another anesthesiologist blinded to the envelops coding. No IM injections will be administered during the perioperative period.

Two days before surgery, patients will visit the outpatient clinic for assessment and explanation about the study protocol. Laboratory investigations will be performed and patients will be informed that they can stop participation in the study at any time without any loss of service.

Inside the operating room, standard monitoring (electrocardiogram, non-invasive blood pressure, heart rate, peripheral oxygen saturation) will be attached and the preliminary values will be recorded. An intravenous cannula 18G will be inserted in the dorsum of the non-dominant hand. Anesthesia will be induced with fentanyl 1 mcg/kg, propofol 1.5-2.0 mg/kg and succinylcholine 1.5 mg/kg.

The intensity of fasciculations will be assessed by an anesthesiologist blinded to the patient's group allotment based on a four-point scale: (0) Absent, (1) Mild: fine fasciculations at the eyes, neck, face or fingers without limb movement, (2) Moderate: fasciculations occurring bilaterally or obvious limb movement and (3) Severe: widespread, sustained fasciculations. After end of fasciculations, the values of heart rate, non-invasive blood pressure and oxygen saturation will be measured and recorded.

Patients will be intubated with an appropriate size cuffed endotracheal tube under direct laryngoscopy after complete muscular relaxation. The endotracheal tube then will be fixed at the appropriate length, by adhesive tape at the angle of the mouth. After 5 minutes of tracheal intubation, the previous values will be recorded again. Subsequent values will be recorded every 5 minutes throughout the surgical procedure. Anesthesia will be maintained with oxygen 100% and sevoflurane (2-3 MAC). Atracurium bromide 0.5 mg/kg will be given after endotracheal intubation. The respiratory tidal volume will be adjusted to keep end-tidal CO2 at 35-40 mmHg. All surgical procedures will be completed by the same surgeon.

At the end of the procedure, sevoflurane will be discontinued; residual neuromuscular blocking agents will be pharmacologically reversed with the standard reversal doses of neostigmine bromide 0.05 mg/kg in atropine sulphate 0.02 mg/kg. The patients then will be ventilated by 100% oxygen till full consciousness regains and the patients start following verbal commands. At that point endotracheal tubes will be removed after gentle suction of secretions through the tube and the oropharyngeal cavity. After the desired spontaneous ventilation, the patients will be shifted to post-anesthesia care unit (PACU).

In PACU, Postoperative care will be standardized for all patients. Pain related to surgical intervention will be treated with paracetamol 1g intravenously (perfalgan; Bristol-Myers Squibb, New York, USA) given every 8h in both group. The total dose of analgesic requirement in the first 24 hours will be recorded. After meeting the discharge criteria, the patients will be discharged to be taken home and cared for, by a responsible adult.

The incidence and severity of myalgia in all patients will be determined 24 hours after surgery by an anesthesiologist who is unaware of the grouping. Myalgia is defined as "a pain with no surgical interference" and is graded based on a four-point scale as follows: (0) no muscle pain, (1) muscle stiffness limited to one area of the body, (2) muscle pain or stiffness noticed spontaneously by a patient who requires analgesics, and (3) incapacitating generalized, severe muscle stiffness or pain.

The postoperative sedation level will be assessed by the Ramsay sedation score which consists of the following six grades: (1) anxious and agitated, (2) cooperative, oriented and tranquil, (3) responding to commands only, (4) brisk response to light glabellar tap or loud auditory stimulus, (5) sluggish response to light glabellar tap or loud auditory stimulus, and (6) no response to light glabellar tap.

Any complications like postoperative nausea, vomiting, dizziness, somnolence, vertigo, confusion will be recorded and managed accordingly. Nausea will be treated by 10 mg metoclopramide intravenously, vomiting will be treated by 4 mg ondansetron intravenously.

Patients' Satisfaction: assessment of patients' satisfaction with the overall preoperative care will be recorded and analyzed.

Statistical analysis:

Data will be performed using a standard SPSS software package version 21 (SPSS Inc., Chicago, Illinois, USA). Data will be expressed as mean ± SD, numbers (n), and median (range). The demographic data will be analyzed by Student t-test. Male and female data will be analyzed with the Chi square test. The consumption of analgesia and sedation in groups will be analyzed by using Student t-test. The incidence and severity of fasciculation and POM will be analyzed using Fisher's exact test. Pearson's r correlation will be used to test the correlation between fasciculations and postoperative myalgia. A p-value of <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* age 20-60 years
* either sex
* ASA physical status I or II

Exclusion Criteria:

* known allergy to duloxetine, abnormal renal and liver function tests, history of chronic pain
* regular medication with SNRI or analgesics (excluding acetaminophen and nonsteroidal anti-inflammatory drugs)
* patients with a history of seizure disorders
* hyperkalemia
* systemic illness like hypertension
* diabetes
* increased intracranial and intraocular pressure
* pregnant or breast-feeding females.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Four-point scale for myalgia | 24 hours
  Myalgia is defined as "a pain with no surgical interference"

SECONDARY OUTCOMES:
Four-point scale for fasciculations | 5 minutes
  Score to assess the intensity of fasciculations
Ramsay sedation score | 24 hours
  To assess the postoperative sedation level
Postoperative Complications | 24 hours
  Percentage of patients with any complications will be recorded and treated

CONTACTS AND LOCATIONS:
Overall Officials: OSAMA A. IBRAHIM, MD, Study Chair — Assiut University
Locations (1):
- Assiut university hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided